CLINICAL TRIAL: NCT05172375
Title: Development of a Model for Shared Care in the Interface Between General Practice and Mental Health Care - a Co-production Study
Brief Title: Development of a Model for Shared Care in the Interface Between General Practice and Mental Health Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Michael Haurum Marcussen, Dr., Psychiatric Research Unit, Region Zealand, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRURegionZealand3
Record Dates: First submitted 2021-11-11; First posted 2021-12-29 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Anxiety Disorders; Depressive Disorder
Keywords: Shared care; Mental Health services; General practice; Mental health recovery; Well-being
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: The study is designed as a non-randomized intervention study with pre- and post design and with a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Shared Care model - intervention group (Experimental): The patients are referred to outpatient clinics based on their home address. The two outpatient clinics should be comparable in terms of patients' diagnoses and staffing. The Shared Care model consists of the following key elements: Shared care is a collaboration between general practice and mental health services and enables a 'best of both worlds' scenario with the opportunity to provide holistic care of high quality to support the recovery process of people with mental health difficulties. The final version of the intervention can only be determined based on the results of the research steps 1+2.
  Interventions: Behavioral: Shared Care Model
- Treatment as usual - Control group (No Intervention): The patients are referred to outpatient clinics based on their home address. The two outpatient clinics should be comparable in terms of patients' diagnoses and staffing. In the control group the patients will receive treatment as usual.

INTERVENTIONS:
Behavioral: Shared Care Model — The Shared Care model consists of the following key elements: Shared care is a collaboration between general practice and mental health services and enables a 'best of both worlds' scenario with the opportunity to provide holistic care of high quality to support the recovery process of people with mental health difficulties.
  Arms: The Shared Care model - intervention group

SUMMARY:
Recent research has underlined that mental health of people with depression and anxiety has deteriorated over the last decades in Denmark as well as internationally, and has reached a degree where it is perceived as a global health challenge. By now, depression is the most common reason for early retirement on health grounds in Denmark. Early intervention in relation to patients with depression and anxiety is essential, as research further shows that many young people with mental health difficulties drop out of education and work. The overall purpose is to develop a shared care intervention in co-production with users, and to increase their recovery by strengthening the support and treatment using a newly developed shared care model.

The study is designed as a non-randomized intervention study with a control group. Comparative analyzes will be performed with pre- and post-assessments. Patients will be recruited between August 2022 and February 2023. The patients are referred to outpatient clinics based on their home address. The two outpatient clinics should be comparable in terms of patients' diagnoses and staffing. ward. Mental health status and well-being are the primary outcomes. Self-reported questionnaires will be administered to both groups before and after the intervention.

The study will be approved by the Research Ethical Committee of University of Southern Denmark and Region Zealand. The study findings will be published in peer-reviewed journals and presented at national and international conferences.

DETAILED DESCRIPTION:
Background Recent research has underlined that mental health of people with depression and anxiety has deteriorated over the last decades in Denmark as well as internationally, and has reached a degree where it is perceived as a global health challenge. Depression and anxiety affect individuals' psychosocial well-being and occupational functioning and are increasing causes of sick leave in high-income countries. By now, depression is the most common reason for early retirement on health grounds in Denmark. Early intervention in relation to patients with depression and anxiety is essential, as research further shows that many young people with mental health difficulties drop out of education and work. Yet it appears that people with mental health difficulties do not receive adequate and sufficient support and treatment. Even though Shared Care between general practice and mental health service was initiated in Denmark more than 10 years ago, the collaboration between the two sectors continues to be challenged. Nonetheless, general practice remains central for the course of treatment of anxiety and depression as the majority of people with these disorders are diagnosed and treated in the primary sector. Among international researchers, there is consensus that most patients should continue to be treated in general practice, however the treatment could be optimized through strengthened collaboration between general practice and mental healthcare services. There is an increasing recognition that improving the treatment and outcomes for people with mental health problems requires service models that integrate mental healthcare within primary healthcare practice. Shared care enables a 'best of both worlds' scenario with the opportunity to provide holistic care of high quality to support the recovery process of people with mental health difficulties. Shared care should lead to pooling of expertise and enhanced creativity in problem-solving. It should also decrease the number of patients 'left in limbo' between primary and secondary sector, with patients and carers feeling that they are failing to make progress through the healthcare system. The most recent Cochrane systematic review of the evidence base for shared care (2013) concluded that shared care interventions significantly improve treatment outcomes compared to treatment as usual. In a situation where researchers, patients and policymakers continue to push for the adoption of shared care between general practice and mental health service, and bearing in mind that the most recent review is almost ten years old, we find that a systematic review of recent studies of shared care is timely, notably to provide a synthesis of the best available evidence for recommendations for future shared care interventions. There is also a great desire for a high degree of user involvement in the project, partly for the purpose of learning for all parties involved, and furthermore to strengthen implementation. Involving users in the study will enhance our understanding of stakeholders' perspectives in relation to their support, treatment, and recovery process. However, there is a lack of stakeholder involvement in this type of research. The project follows Psychiatry in Region Zealand's overall strategy for implementing Recovery, on the assumption that a shared cared approach strengthens the treatment and the social support, and thereby supports the recovery process of people with mental illness. The overall purpose is to develop a shared care intervention in co-production with users, and to increase their recovery by strengthening the support and treatment using a newly developed shared care model.

Methods A systematic review (Step 1) is followed by an explanatory study (Step 2) with interviews of relevant stakeholders in shared care to explore how general practitioners, mental health staff and patients perceive collaboration, user involvement and the course of treatment in shared care. Both steps are planned to inform and qualify an intervention (Step 3). It is the assumption that the involvement of patients in all phases will result in a higher relevance for both clinical practice and patients (ref.). Therefore, we have decided to create a new Shared Care intervention that will be developed in co-production with the users. Co-production in research is defined as "an approach in which researchers, practitioners and the public work together, sharing power and responsibility from the start to the end of the project, including the generation of knowledge." (NIHR 2021).

Step 1 - Systematic review A systematic review is conducted based on the following research questions 1) What characterizes a shared care model? 2) how do general practitioners, mental health providers, and patients experience shared care? The review is planned and will be implemented and published based on PRISMA guidelines. We will conduct a search in the following databases: Medline, CINAHL, PsychINFO and EMBASE for both qualitative and quantitative studies, published in the period January 2001 to January 2022. Two independent researchers will conduct screening on both title and abstract level (MM and BN). Furthermore, full-text reading and quality assessment (risk of bias) will be based on CASP checklists. The project is registered in Prospero (287989) and carried out through the software platform covidence.org.

Step 2 - Perspectives on shared care This study is intended to supplement Step 1 (systematic review) with a user perspective (both people with mental illness and health professionals) on shared care. Phase 2 will be an exploratory study based on interviews with people involved in shared care in Region Zealand, general practitioners, patients, as well as health professionals from the mental health service. The interviews will be conducted to investigate what people with mental illness and health professionals find important in the pathways as well as their perspectives on shared care, collaboration, and recovery. Informants will be found with a view to maximal variation in terms of age, sex, profession, diagnosis, and duration of illness. A semi-structured interview guide will be prepared and data analysis will be based on thematic analysis, inspired by Kvale & Brinkmann and Coffey & Atkinson.

This study is based on the two previous steps, including a systematic review (ID: 287989) and an exploration of users' experiences of shared care - collaboration between general practice and mental healthcare. Both steps are planned to inform and qualify the intervention but no further described in this protocol.

Study design The study is designed as a non-randomized intervention study with a control group. Comparative analyzes will be performed with pre- and post-assessments. Patients will be recruited between August 2022 and February 2023. The patients are referred to outpatient clinics based on their home address. The two outpatient clinics should be comparable in terms of patients' diagnoses and staffing. The trial is registered in ClinicalTrials.gov (NCT not yet assigned) and adhered to the Consort guidelines.

Intervention The Shared Care model consists of the following key elements: Shared care is a collaboration between general practice and mental health services and enables a 'best of both worlds' scenario with the opportunity to provide holistic care of high quality to support the recovery process of people with mental health difficulties. The final version of the intervention can only be determined based on the results of the research steps 1+2.

Study population The participants are adults aged 18 - 65 years, diagnosed with depression and anxiety, and referred to outpatient clinics in Region Zealand.

Procedure for recruitment Data collection via questionnaires, which will be administered to the patients at the first visit in the outpatient clinic and after 3 months. Patients who did not consent to participation or failed to complete the questionnaire at the first visit in the outpatient-clinic were excluded from the study.

Primary outcome Mental health status is valid and reliable indicator of the patients self-reported mental state and well-being. Mental status is assessed using the standardized Short Form Health Survey (SF-36), first developed in the US by Ware and Sherbourne. A Danish translation of the original English-language version will be used.

Secondary outcomes The patients level of function is assessed using the Global assessment of functioning (GAF), and their satisfaction is measured with the client satisfaction score scale (CSQ-8) and the quality of Life enjoyment and satisfaction questionnaire (Q-LES-Q (SF). The patients' recovery will be assessed by the 24-item recovery assessment scale-revised (RAS-R). All scales have been validated in a Danish population. The implementation of the Shared Care model will be ensured by fidelity assessments. Checklists will be used to ensure that the collaborative meetings are held as planned.

Sample size The sample size calculation is based on an intervention study with SF-36 as the primary outcome, also conducted in Mental health services. In this study, there is a clinically relevant effect size 0.5 with a power 80 ((α = 0.05). Based on this study's sample size calculation, 120 patients in each group are needed (intervention and control).

Ethical considerations Information of participants and data management will be planned in accordance with the Helsinki Declaration. Informed consent based on information, both written and verbally, about the aim, purpose and use of the study and the data collection will be obtained from all participants. Furthermore, all participants will be informed that their participation was voluntary, that they could withdraw their consent at any time without consequences, and that their statements would be treated confidentially and anonymized. Data will be entered into the EasyTrial © Online Clinical Trial Management system. All personal identifiers will be removed or disguised during analysis to preclude personal identification. The project will be reported to the Danish Data Protection Agency and the Region Zealand Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Out patient
* Diagnosed with: Anxiety and Depression
* Aged 18 - 65 years

Exclusion Criteria:

* Cognitive deficit
* Patients who did not consent to participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Mental Health Status | At baseline and after 3 months
  Mental health status is valid and reliable indicator of the patients self-reported mental state and well-being. Mental status is assessed using the standardized Short Form Health Survey (SF-36). Its 36 items are grouped into eight domains. The summed scores for each of the eight domains were plotted on a scale from 0 (worst) to 100 (best), with higher scores indicating better health
Change in mental health recovery | Baseline and after 3 months.
  The patients' recovery will be assessed by the 24-item recovery assessment scale-revised (RAS-R) - a questionnaire. It is a self-report instrument measuring mental health recovery. The RAS-R thus consists of 24 items on five-level scales. These items can be added up to produce summary scales representing five dimensions of personal recovery.

SECONDARY OUTCOMES:
Change in level of function | Baseline and after 3 months.
  The patients level of function is assessed using the Global assessment of functioning (GAF) - a questionnaire. The GAF is a scale from 0 to 100 where higher scores indicate greater levels of functioning.
Change in Patient Satisfaction | Baseline and after 3 months.
  Satisfaction is measured with the client satisfaction score scale (CSQ-8) - a questionnaire.
  * For overall score, sum item responses, range from 8-32, higher score indicates higher satisfaction.
Change in Patient Satisfaction | Baseline and after 3 months.
  The Quality-of-Life Enjoyment and Satisfaction Questionnaire.
Improvement in collaboration between general practice and mental health | Baseline and after 3 months.
  The Collaborative Practice Scale.
Improvement in collaboration between general practice and mental health | Baseline and after 3 months.
  Shared Decision-Making Questionnaire (SDM-Q9).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marcussen, Dr., Principal Investigator — University of Southern Denmark (SDU), Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Christensen TN, Wallstrom IG, Bojesen AB, Nordentoft M, Eplov LF. Predictors of work and education among people with severe mental illness who participated in the Danish individual placement and support study: findings from a randomized clinical trial. Soc Psychiatry Psychiatr Epidemiol. 2021 Sep;56(9):1669-1677. doi: 10.1007/s00127-021-02107-8. Epub 2021 May 25. PMID 34032866
- [Result] Mojtabai R, Olfson M, Han B. National Trends in the Prevalence and Treatment of Depression in Adolescents and Young Adults. Pediatrics. 2016 Dec;138(6):e20161878. doi: 10.1542/peds.2016-1878. Epub 2016 Nov 14. PMID 27940701
- [Result] Kennedy N, Foy K, Sherazi R, McDonough M, McKeon P. Long-term social functioning after depression treated by psychiatrists: a review. Bipolar Disord. 2007 Feb-Mar;9(1-2):25-37. doi: 10.1111/j.1399-5618.2007.00326.x. PMID 17391347
- [Result] Iancu SC, Batelaan NM, Zweekhorst MB, Bunders JF, Veltman DJ, Penninx BW, van Balkom AJ. Trajectories of functioning after remission from anxiety disorders: 2-year course and outcome predictors. Psychol Med. 2014 Feb;44(3):593-605. doi: 10.1017/S0033291713001050. Epub 2013 May 10. PMID 23659543
- [Result] Rugulies R, Aust B. Work and mental health: what do we know and how can we intervene? Scand J Work Environ Health. 2019 Nov 1;45(6):529-532. doi: 10.5271/sjweh.3856. Epub 2019 Oct 16. No abstract available. PMID 31616953
- [Result] Sogaard HJ, Bech P. Psychiatric disorders in long-term sickness absence -- a population-based cross-sectional study. Scand J Public Health. 2009 Sep;37(7):682-9. doi: 10.1177/1403494809344357. Epub 2009 Aug 21. PMID 19700479
- [Result] Manthey TJ, Goscha R, Rapp C. Barriers to supported education implementation: implications for administrators and policy makers. Adm Policy Ment Health. 2015 May;42(3):245-51. doi: 10.1007/s10488-014-0583-z. PMID 25145926
- [Result] Ringeisen H, Langer Ellison M, Ryder-Burge A, Biebel K, Alikhan S, Jones E. Supported education for individuals with psychiatric disabilities: State of the practice and policy implications. Psychiatr Rehabil J. 2017 Jun;40(2):197-206. doi: 10.1037/prj0000233. Epub 2017 Feb 9. PMID 28182470
- [Result] Hunt J, Eisenberg D. Mental health problems and help-seeking behavior among college students. J Adolesc Health. 2010 Jan;46(1):3-10. doi: 10.1016/j.jadohealth.2009.08.008. Epub 2009 Oct 20. PMID 20123251
- [Result] Weitkamp K, Klein E, Midgley N. The Experience of Depression: A Qualitative Study of Adolescents With Depression Entering Psychotherapy. Glob Qual Nurs Res. 2016 May 16;3:2333393616649548. doi: 10.1177/2333393616649548. eCollection 2016 Jan-Dec. PMID 28462338
- [Result] Bauer J, Okkels N, Munk-Jorgensen P. State of psychiatry in Denmark. Int Rev Psychiatry. 2012 Aug;24(4):295-300. doi: 10.3109/09540261.2012.692321. PMID 22950767
- [Derived] Marcussen M, Berring L, Horder M, Sondergaard J, Norgaard B. Development of a model for shared care between general practice and mental healthcare: a protocol for a co-production study. BMJ Open. 2022 Oct 31;12(10):e061575. doi: 10.1136/bmjopen-2022-061575. PMID 36316081